CLINICAL TRIAL: NCT00513292
Title: A Randomized Phase III Trial Comparing a Neoadjuvant Regimen of FEC-75 Followed by Paclitaxel Plus Trastuzumab With a Neoadjuvant Regimen of Paclitaxel Plus Trastuzumab Followed by FEC-75 Plus Trastuzumab in Patients With HER-2 Positive Operable Breast Cancer
Brief Title: Combination Chemotherapy and Paclitaxel Plus Trastuzumab in Treating Women With Palpable Breast Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00341; NCI-2009-00341 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000559039; ACOSOG-Z1041; Z1041 (Other: American College of Surgeons Oncology Group); ACOSOG-Z1041 (Other: CTEP); U10CA012027 (NIH)
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Results first posted 2015-09-29 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: HER2/Neu Positive; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Epirubicin; Paclitaxel; Taxes; Trastuzumab; PF-05280014

ARMS (2):
- FEC-75 then Paclitaxel/trastuzumab (Active Comparator): Patients receive FEC comprising fluoroucacil IV, epirubicin hydrochloride IV, and cyclophosphamide IV on day 1. Treatment repeats every 21 days for 4 courses. Beginning 21 days after completion of FEC, patients receive paclitaxel IV once weekly and trastuzumab (Herceptin) IV once weekly for 12 weeks. Within 6 weeks after completion of paclitaxel and trastuzumab, patients undergo surgery. Beginning 3-4 weeks after surgery, patients receive trastuzumab IV once every 3 weeks for up to 52 weeks.
  Interventions: Drug: Cyclophosphamide; Drug: Epirubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Procedure: Therapeutic Conventional Surgery; Biological: Trastuzumab
- Paclitaxel/trastuzumab then trastuzumab/FEC-75 (Experimental): Patients receive paclitaxel IV once weekly and trastuzumab IV once weekly for 12 weeks. Beginning 7 days after the completion of paclitaxel and trastuzumab, patients receive FEC comprising fluoroucacil IV, epirubicin IV, and cyclophosphamide IV on day 1. Treatment repeats every 21 days for 4 courses. Patients also receive trastuzumab IV once weekly for an additional 12 weeks. Within 6 weeks after completion of FEC and trastuzumab, patients undergo surgery. Beginning 3-4 weeks after surgery, patients receive trastuzumab as in arm I.
  Interventions: Drug: Cyclophosphamide; Drug: Epirubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Procedure: Therapeutic Conventional Surgery; Biological: Trastuzumab

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Epirubicin Hydrochloride — Given IV
  Other Names: Ellence; IMI-28; Pharmorubicin PFS
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Procedure: Therapeutic Conventional Surgery — Undergo surgery
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; PF-05280014; rhuMAb HER2; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar PF-05280014

SUMMARY:
This randomized phase III trial is studying giving fluorouracil together with epirubicin and cyclophosphamide followed by paclitaxel and trastuzumab to see how well it works compared with giving paclitaxel together with trastuzumab followed by fluorouracil, epirubicin, cyclophosphamide, and trastuzumab in treating women with palpable breast cancer that can be removed by surgery. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether it is more effective to give combination chemotherapy before or after treatment with paclitaxel plus trastuzumab.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary objective of this study is to compare the pathologic complete response rate (pCR) within the breast of a sequential regimen of concurrent weekly paclitaxel and trastuzumab, followed by continued weekly trastuzumab administered concurrently with FEC-75 (Arm 2), to the pCR rate of a sequential regimen of FEC-75 alone followed by concurrent weekly paclitaxel and trastuzumab (Arm 1).

SECONDARY OBJECTIVES:

I. To estimate the cardiotoxicity of a sequential regimen of concurrent weekly paclitaxel and trastuzumab, followed by continued weekly trastuzumab administered concurrently with FEC-75, followed postoperatively by q 3 week trastuzumab for a total duration of trastuzumab therapy through 52 weeks from the first dose (Arm 2), and compare the cardiotoxicity to that of a sequential regimen of FEC-75 alone followed by concurrent weekly paclitaxel and trastuzumab, followed by q 3 week trastuzumab for a total duration of trastuzumab therapy through 52 weeks from the first dose (Arm 1).

II. To compare the combined pCR rate in the breast and ipsilateral axilla obtained with the two regimens evaluated in this study.

III. To compare the clinical response rates (cRR) of the two regimens evaluated in this study.

IV. To compare the non-cardiac toxicity of the two regimens evaluated in this study.

V. To compare breast conservation rates achieved with the two regimens evaluated in this study.

VI. To evaluate disease-free survival and overall survival at 5 years post-randomization.

VII. To correlate pCR rate with potential molecular markers of response.

OUTLINE: Patients are stratified by clinical tumor size (breast tumor size < 2 cm and nodal metastases < 2 cm vs breast tumor size < 2 cm and nodal metastases ≥ 2 cm vs breast tumor size 2-4 cm [any nodal status] vs breast tumor size ≥ 4 cm [any nodal status]), age (< 50 vs ≥ 50) and hormone receptor status (estrogen receptor [ER]- and progesterone receptor [PgR]-negative vs ER- and/or PgR-positive). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive FEC comprising fluoroucacil intravenously (IV), epirubicin hydrochloride IV, and cyclophosphamide IV on day 1. Treatment repeats every 21 days for 4 courses. Beginning 21 days after completion of FEC, patients receive paclitaxel IV once weekly and trastuzumab (Herceptin) IV once weekly for 12 weeks. Within 6 weeks after completion of paclitaxel and trastuzumab, patients undergo surgery. Beginning 3-4 weeks after surgery, patients receive trastuzumab IV once every 3 weeks for up to 52 weeks.

ARM II: Patients receive paclitaxel IV once weekly and trastuzumab IV once weekly for 12 weeks. Beginning 7 days after completion of paclitaxel and trastuzumab, patients receive FEC comprising fluoroucacil IV, epirubicin IV, and cyclophosphamide IV on day 1. Treatment repeats every 21 days for 4 courses. Patients also receive trastuzumab IV once weekly for an additional 12 weeks. Within 6 weeks after completion of FEC and trastuzumab, patients undergo surgery. Beginning 3-4 weeks after surgery, patients receive trastuzumab as in arm I.

After completion of study therapy, patients are followed every 3 months for 1 year and then every 6 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of invasive adenocarcinoma by core needle biopsy

  * Fine needle aspiration allowed provided primary tumor size < 2 cm and lymph node metastases are present
  * Excisional biopsy of the primary tumor allowed provided biopsy-positive lymph nodes are present
* Primary tumor ≥ 2 cm and/or ≥ 1 biopsy-positive lymph node
* HER2-positive disease

  * Confirmation by fluorescent in situ hybridization (FISH) requires gene amplification
  * Confirmation by immunohistochemistry (IHC) requires a strongly positive (3+) staining intensity score
* Ductal carcinoma in situ (DCIS) or synchronous DCIS of the contralateral breast regardless of prior therapy allowed

  * Synchronous invasive breast cancer not allowed
* Ipsilateral DCIS treated by local excision with or without hormonal therapy allowed

  * Those treated with radiation therapy are not allowed
* No definitive clinical or radiologic evidence of metastatic disease
* No history of invasive breast cancer
* Hormone receptor status known
* Menopausal status not specified
* ECOG performance status of 0 -1
* Absolute neutrophil count ≥ 1,200/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin normal unless the patient has a grade 1 bilirubin elevation (normal to 1.5 times upper limit of normal [ULN]) resulting from Gilbert disease or similar syndrome due to slow conjugation of bilirubin
* Alkaline phosphatase ≤ 2.5 times ULN
* AST ≤ 1.5 times ULN
* Creatinine normal
* Left ventricular ejection fraction (LVEF) ≥ 55 by multi gated acquisition scan (MUGA) or echocardiogram (ECHO) within the past 3 months
* Patients with either skeletal pain or alkaline phosphatase that is > ULN but ≤ 2.5 times ULN allowed if bone scans fail to demonstrate metastatic disease

  * Suspicious findings on bone scan must be confirmed as benign by x-ray, MRI, or biopsy
* Prior non-breast malignancies allowed if disease-free for 5 years since completion of initial treatment regimen and deemed by their physician to be at low risk for recurrence

  * Patients who had the following cancers are eligible if diagnosed and treated within the past 5 years:

    * Carcinoma in situ of the cervix
    * Colon carcinoma in situ
    * Melanoma in situ
    * Basal cell and squamous cell carcinoma of the skin
* No cardiac disease that would preclude the use of epirubicin hydrochloride or trastuzumab (Herceptin®) including any of the following:

  * Active cardiac disease
  * Angina pectoris that requires the use of antianginal medication
  * Cardiac arrhythmia requiring medication
  * Severe conduction abnormality
  * Clinically significant valvular disease
  * Cardiomegaly on chest x-ray
  * Ventricular hypertrophy on EKG
  * Patient's with poorly controlled hypertension ( i.e., diastolic greater than 100 mm/Hg)

    * Patients with hypertension that is well controlled on medication are eligible
  * History of cardiac disease
  * Myocardial infarction documented as a clinical diagnosis or by EKG or any other tests
  * Documented congestive heart failure
  * Documented cardiomyopathy
* No sensory or motor neuropathy ≥ grade 2, as defined by the NCI's CTCAE v3.0
* Women of reproductive potential must agree to use an effective non-hormonal method of contraception during therapy
* Women of child bearing potential must have a negative urine or serum pregnancy test within 2 weeks of registration
* Not pregnant or nursing
* No psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements
* No non-malignant systemic disease (e.g., cardiovascular, renal, hepatic) that would preclude treatment with either of the treatment regimens
* No prior surgical axillary staging procedure

  * Prior non-excisional biopsy of an axillary node allowed
* No prior treatment for this breast cancer

  * Hormonal therapy allowed if had been given for up to a total of 28 days anytime after diagnosis and before study entry
  * Hormonal therapy must stop at or before study entry and be re-started, if indicated, following surgery
* No prior therapy with anthracyclines or taxanes for any malignancy
* No other investigational agents within the past 30 days
* No concurrent sex hormonal therapy (e.g., birth control pills, ovarian hormonal replacement therapy)
* No concurrent therapy with any hormonal agent such as raloxifene, tamoxifen, or other selective estrogen receptor modulator (SERM), either for osteoporosis or breast cancer prevention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2007-07; Primary Completion 2012-06 (Actual); Study Completion 2013-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aman Buzdar, Principal Investigator — American College of Surgeons
Locations (115):
- United States (114):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Eden Hospital Medical Center, Castro Valley, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Saint Rose Hospital, Hayward, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Morton Plant Hospital, Clearwater, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Presence Resurrection Medical Center, Chicago, Illinois
  - Saint Francis Hospital and Health Centers, Beech Grove, Indiana
  - Franciscan Saint Francis Health-Indianapolis, Indianapolis, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Unspecified Site, Rockville, Maryland
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Singing River Hospital, Pascagoula, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - UMDNJ - New Jersey Medical School, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Orange Regional Medical Center, Middletown, New York
  - MidHudson Regional Hospital of Westchester Medical Center, Poughkeepsie, New York
  - Staten Island University Hospital, Staten Island, New York
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Veteran Affairs Medical Center, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Nashville Breast Center, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Zale Lipshy University Hospital, Dallas, Texas
  - Clements University Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Danville Regional Medical Center, Danville, Virginia
  - Sentara Port Warwick, Newport News, Virginia
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Oconomowoc Memorial Hospital-ProHealth Care Inc, Oconomowoc, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- San Juan City Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Buzdar AU, Suman VJ, Meric-Bernstam F, Leitch AM, Ellis MJ, Boughey JC, Unzeitig GW, Royce ME, Hunt KK. Disease-Free and Overall Survival Among Patients With Operable HER2-Positive Breast Cancer Treated With Sequential vs Concurrent Chemotherapy: The ACOSOG Z1041 (Alliance) Randomized Clinical Trial. JAMA Oncol. 2019 Jan 1;5(1):45-50. doi: 10.1001/jamaoncol.2018.3691. PMID 30193295
- [Derived] Lesurf R, Griffith OL, Griffith M, Hundal J, Trani L, Watson MA, Aft R, Ellis MJ, Ota D, Suman VJ, Meric-Bernstam F, Leitch AM, Boughey JC, Unzeitig G, Buzdar AU, Hunt KK, Mardis ER. Genomic characterization of HER2-positive breast cancer and response to neoadjuvant trastuzumab and chemotherapy-results from the ACOSOG Z1041 (Alliance) trial. Ann Oncol. 2017 May 1;28(5):1070-1077. doi: 10.1093/annonc/mdx048. PMID 28453704
- [Derived] Buzdar AU, Suman VJ, Meric-Bernstam F, Leitch AM, Ellis MJ, Boughey JC, Unzeitig G, Royce M, McCall LM, Ewer MS, Hunt KK; American College of Surgeons Oncology Group investigators. Fluorouracil, epirubicin, and cyclophosphamide (FEC-75) followed by paclitaxel plus trastuzumab versus paclitaxel plus trastuzumab followed by FEC-75 plus trastuzumab as neoadjuvant treatment for patients with HER2-positive breast cancer (Z1041): a randomised, controlled, phase 3 trial. Lancet Oncol. 2013 Dec;14(13):1317-25. doi: 10.1016/S1470-2045(13)70502-3. Epub 2013 Nov 13. PMID 24239210

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total Enrolled: 282, 2 patients withdrew consent before starting treatment, 280 patients started the treatment and are eligible for primary analysis.
Groups:
- FEC-75 Then Paclitaxel/Trastuzumab: Patients receive FEC comprising fluorouracil IV, epirubicin hydrochloride IV, and cyclophosphamide IV on day 1. Treatment repeats every 21 days for 4 courses. Beginning 21 days after completion of FEC, patients receive paclitaxel IV once weekly and trastuzumab (Herceptin) IV once weekly for 12 weeks. Within 6 weeks after completion of paclitaxel and trastuzumab, patients undergo surgery. Beginning 3-4 weeks after surgery, patients receive trastuzumab IV once every 3 weeks for up to 52 weeks. epirubicin hydrochloride: Given IV, cyclophosphamide: Given IV, paclitaxel: Given IV, trastuzumab: Given IV, therapeutic conventional surgery: Undergo surgery, laboratory biomarker analysis: Correlative studies
- Paclitaxel/Trastuzumab Then Trastuzumab/FEC-75: Patients receive paclitaxel IV once weekly and trastuzumab IV once weekly for 12 weeks. Beginning 7 days after the completion of paclitaxel and trastuzumab, patients receive FEC comprising fluorouracil IV, epirubicin IV, and cyclophosphamide IV on day 1. Treatment repeats every 21 days for 4 courses. Patients also receive trastuzumab IV once weekly for an additional 12 weeks. Within 6 weeks after completion of FEC and trastuzumab, patients undergo surgery. Beginning 3-4 weeks after surgery, patients receive trastuzumab as in arm I. epirubicin hydrochloride: Given IV, cyclophosphamide: Given IV, paclitaxel: Given IV, trastuzumab: Given IV, therapeutic conventional surgery: Undergo surgery, laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | FEC-75 Then Paclitaxel/Trastuzumab | Paclitaxel/Trastuzumab Then Trastuzumab/FEC-75
Started | 138 | 142
Completed | 138 | 142
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total enrolled: 282, 2 withdrew consent before start of treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | FEC-75 Then Paclitaxel/Trastuzumab | Paclitaxel/Trastuzumab Then Trastuzumab/FEC-75 | Total
Number analyzed (Participants) | 138 | 142 | 280
Age, Continuous [Median (Full Range); unit: years] | 51 [32 to 76] | 48 [28 to 73] | 50 [28 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 142 | 280
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 138 | 142 | 280

OUTCOME MEASURES:

1. Primary Outcome: pCR Within the Breast, Defined as no Evidence of Invasive Tumor Remaining in the Breast at Surgery Following Completion of Chemotherapy
Description: Pathological complete response (pCR) rates will be based on institutional pathology reports. In the final analysis for publication, rates will be based on blinded central review of these institutional pathology reports. The Chi-squared test will be conducted at the two-sided 0.05 level. A 95% confidence interval will be computed for the difference in pCR rates.
Time Frame: Up to 5 years
Population: All patients who started study treatment are included in the analysis of the primary endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- FEC-75 Then Paclitaxel/Trastuzumab: Patients receive Fluorouracil, epirubicin, and cyclophosphamide (FEC) comprising fluorouracil IV, epirubicin hydrochloride IV, and cyclophosphamide IV on day 1. Treatment repeats every 21 days for 4 courses. Beginning 21 days after completion of FEC, patients receive paclitaxel IV once weekly and trastuzumab (Herceptin) IV once weekly for 12 weeks. Within 6 weeks after completion of paclitaxel and trastuzumab, patients undergo surgery. Beginning 3-4 weeks after surgery, patients receive trastuzumab IV once every 3 weeks for up to 52 weeks. epirubicin hydrochloride: Given IV, cyclophosphamide: Given IV, paclitaxel: Given IV, trastuzumab: Given IV, therapeutic conventional surgery: Undergo surgery, laboratory biomarker analysis: Correlative studies
Arm/Group | FEC-75 Then Paclitaxel/Trastuzumab | Paclitaxel/Trastuzumab Then Trastuzumab/FEC-75
Number analyzed (Participants) | 138 | 142
percentage of participants | 56.5 [47.8 to 64.9] | 54.2 [45.7 to 62.6]
Statistical Analysis 1: Comparison: FEC-75 Then Paclitaxel/Trastuzumab vs Paclitaxel/Trastuzumab Then Trastuzumab/FEC-75; The difference in pCR rates between treatment arms for pCR within the Breast, Defined as no Evidence of Invasive Tumor Remaining in the Breast at Surgery Following Completion of Chemotherapy; Test type: Superiority or Other; p = .7, Chi-squared; difference in percentages between arms = 2.3, 95% CI 2-sided [-9.3 to 13.9]

2. Secondary Outcome: Combined pCR Rate in the Breast and Axillary Lymph Nodes Defined as no Evidence of Invasive Tumor Remaining in Either the Breast or Axillary Nodes at Surgery Following Completion of Chemotherapy
Description: pCR Rate in the Breast and Axillary Lymph Nodes Defined as no Evidence of Invasive Tumor Remaining in Either the Breast or Axillary Nodes at Surgery Following Completion of Chemotherapy (among those with Metastasis to movable ipsilateral axillary lymph node(s) (cN1-3) disease).
Time Frame: Up to 5 years
Population: All patients who had clinical N1-3 disease prior to the start of treatment are included in the analysis of the pCR rate in the breast and axillary lymph nodes.
Measure: Number (95% Confidence Interval); unit: Percentage (95% confidence Interval)
Arm/Group | FEC-75 Then Paclitaxel/Trastuzumab | Paclitaxel/Trastuzumab Then Trastuzumab/FEC-75
Number analyzed (Participants) | 89 | 90
Percentage (95% confidence Interval) | 48.3 [37.6 to 59.2] | 46.7 [36.4 to 56.9]

3. Secondary Outcome: Asymptomatic Decreases From Baseline in Left Ventricular Ejection Fraction (LVEF) at Week 12
Description: The summary of asymptomatic decrease in LVEF.
Time Frame: Baseline, at 12 week
Population: All patients who had a MUGA or ECHO performed at week 12 are included in the summary of asymptomatic changed in LVEF at week 12.
Measure: Number; unit: Percentage of participants
Arm/Group | FEC-75 Then Paclitaxel/Trastuzumab | Paclitaxel/Trastuzumab Then Trastuzumab/FEC-75
Number analyzed (Participants) | 130 | 137
Percentage of participants
  no decrease or decrease < 10%, still above LLN | 92.3 | 82.5
  decrease < 10%, below lower limit of normal (LLN) | 0.8 | 0
  decrease 10-15%, still above lower limit of normal | 6.2 | 11.7
  decrease 10-15%, below lower limit of normal (LLN) | 0 | 0
  decrease > 15%, still above lower limit of norm | 0.8 | 2.9
  decrease > 15%, below lower limit of normal | 0 | 2.9

4. Secondary Outcome: Asymptomatic Decreases From Baseline in LVEF at Week 24
Description: The summary of asymptomatic changed in LVEF.
Time Frame: Baseline, at 24 week
Population: All patients who had a MUGA or ECHO performed at week 24 are included in the summary of asymptomatic changed in LVEF at week 24.
Measure: Number; unit: Percentage of Participants
Arm/Group | FEC-75 Then Paclitaxel/Trastuzumab | Paclitaxel/Trastuzumab Then Trastuzumab/FEC-75
Number analyzed (Participants) | 126 | 130
Percentage of Participants
  no decrease or decrease < 10%, still above LLN | 83.3 | 73.1
  decrease < 10%, below lower limit of normal (LLN) | 0.8 | 3.1
  decrease 10-15%, still above lower limit of normal | 7.9 | 15.4
  decrease 10-15%, below lower limit of normal (LLN) | 2.4 | 0.8
  decrease > 15%, still above lower limit of normal | 1.6 | 6.9
  decrease > 15%, below lower limit of normal (LLN) | 4.0 | 0.8

5. Secondary Outcome: LVEFs From Regularly Scheduled Multi Gated Acquisition Scan (MUGA)/Echo Scans as Reported at 12 Week
Description: All patients who had a MUGA or ECHO performed at week 12 are included in the summary of asymptomatic changed in LVEF at week 12. Difference from pretreatment LVEF (%) at 12 weeks [median change from baseline Inter Quartile Range (IQR)].
Time Frame: At 12 week
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | FEC-75 Then Paclitaxel/Trastuzumab | Paclitaxel/Trastuzumab Then Trastuzumab/FEC-75
Number analyzed (Participants) | 130 | 137
percent | 2 [-5 to 2] | -3 [-7 to 0]

6. Secondary Outcome: Change in LVEFs (From Regularly Scheduled Multi Gated Acquisition Scan (MUGA)/Echo Scans) From Baseline and at 24 Week
Description: Difference from pretreatment LVEF (%) at 24 weeks [median change from baseline Inter Quartile Range (IQR)].
Time Frame: Baseline, at 24 week
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | FEC-75 Then Paclitaxel/Trastuzumab | Paclitaxel/Trastuzumab Then Trastuzumab/FEC-75
Number analyzed (Participants) | 126 | 130
percent | -3 [-7 to 0] | -4 [-9 to 0]

7. Secondary Outcome: Breast Conservation
Description: Surgery was categorized as breast conserving surgery ("Partial Mastectomy") or non-conserving surgery ("Total Mastectomy" or "Modified Radical Mastectomy). Reported below is the percentage of patients receiving "Partial Mastectomy". This was calculated by dividing the number of patients receiving "Partial Mastectomy" by the total number of patients undergoing surgery multiplied by 100 (to obtain the percentage).
Time Frame: From time surgery to up to 5 years
Population: All patients that underwent breast surgery were included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | FEC-75 Then Paclitaxel/Trastuzumab | Paclitaxel/Trastuzumab Then Trastuzumab/FEC-75
Number analyzed (Participants) | 130 | 138
percentage of participants | 37.7 | 39.1

8. Secondary Outcome: Disease-free Survival (DFS)
Description: DFS defined as inoperable progressive disease, gross residual disease following definitive surgery, local, regional or distant recurrence, contralateral breast cancer, other second primary cancers, and death prior to recurrence or second primary cancer. DFS of Arm I and Arm II patients will be estimated using the Kaplan-Meier method.
Time Frame: From time to registration to time of event, assessed up to 5 years
Population: All patients that began protocol therapy are included in this analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FEC-75 Then Paclitaxel/Trastuzumab | Paclitaxel/Trastuzumab Then Trastuzumab/FEC-75
Number analyzed (Participants) | 138 | 142
months | NA [NA to NA] — Too few events occurred to report a median and 95% Confidence Interval. | NA [NA to NA] — Too few events occurred to report a median and 95% Confidence Interval.

9. Secondary Outcome: Overall Survival (OS)
Description: OS of Arm I and Arm II patients will be estimated using the Kaplan-Meier method.
Time Frame: From time to registration to death, assessed up to 5 years
Population: All patients that began protocol therapy were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FEC-75 Then Paclitaxel/Trastuzumab | Paclitaxel/Trastuzumab Then Trastuzumab/FEC-75
Number analyzed (Participants) | 138 | 142
months | NA [NA to NA] — Too few events occurred to report a median and 95% Confidence Interval. | NA [NA to NA] — Too few events occurred to report a median and 95% Confidence Interval.

ADVERSE EVENTS:
Groups:
- Arm A: Patients receive FEC comprising fluorouracil IV, epirubicin hydrochloride IV, and cyclophosphamide IV on day 1. Treatment repeats every 21 days for 4 courses. Beginning 21 days after completion of FEC, patients receive paclitaxel IV once weekly and trastuzumab (Herceptin) IV once weekly for 12 weeks. Within 6 weeks after completion of paclitaxel and trastuzumab, patients undergo surgery. Beginning 3-4 weeks after surgery, patients receive trastuzumab IV once every 3 weeks for up to 52 weeks. epirubicin hydrochloride: Given IV, cyclophosphamide: Given IV, paclitaxel: Given IV, trastuzumab: Given IV, therapeutic conventional surgery: Undergo surgery, laboratory biomarker analysis: Correlative studies
- Arm B: Patients receive paclitaxel IV once weekly and trastuzumab IV once weekly for 12 weeks. Beginning 7 days after the completion of paclitaxel and trastuzumab, patients receive FEC comprising fluorouracil IV, epirubicin IV, and cyclophosphamide IV on day 1. Treatment repeats every 21 days for 4 courses. Patients also receive trastuzumab IV once weekly for an additional 12 weeks. Within 6 weeks after completion of FEC and trastuzumab, patients undergo surgery. Beginning 3-4 weeks after surgery, patients receive trastuzumab as in arm I. epirubicin hydrochloride: Given IV, cyclophosphamide: Given IV, paclitaxel: Given IV, trastuzumab: Given IV, therapeutic conventional surgery: Undergo surgery, laboratory biomarker analysis: Correlative studies
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 19/138 | 26/142
Other Adverse Events (participants affected / at risk) | 136/138 | 141/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=138) | Arm B (N=142)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Hemoglobin decreased (Blood and lymphatic system disorders) | 8 (12) | 11 (14)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 3 (3) | 5 (6)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 1 (1)
Eyelid function disorder (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 3 (3)
Anal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 9 (12) | 8 (8)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 4 (6) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (11) | 8 (10)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 6 (6)
Chest pain (General disorders) | 1 (1) | 2 (2)
Chills (General disorders) | 1 (1) | 2 (2)
Edema limbs (General disorders) | 3 (3) | 4 (4)
Fatigue (General disorders) | 13 (23) | 17 (23)
Fever (General disorders) | 6 (7) | 4 (4)
Localized edema (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (2) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 2 (2)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 3 (4)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4)
Skin infection (Infections and infestations) | 5 (5) | 2 (2)
Soft tissue infection (Infections and infestations) | 1 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (7) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 3 (3)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1)
Laboratory test abnormal (Investigations) | 2 (2) | 1 (2)
Leukocyte count decreased (Investigations) | 3 (3) | 8 (12)
Lymphocyte count decreased (Investigations) | 1 (3) | 6 (11)
Neutrophil count decreased (Investigations) | 6 (7) | 13 (20)
Platelet count decreased (Investigations) | 1 (1) | 3 (3)
Serum cholesterol increased (Investigations) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 3 (3)
Weight loss (Investigations) | 3 (4) | 2 (2)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (4) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (4)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Encephalopathy (Nervous system disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 6 (7) | 9 (10)
Neurological disorder NOS (Nervous system disorders) | 1 (9) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (6) | 8 (10)
Syncope (Nervous system disorders) | 2 (2) | 2 (2)
Taste alteration (Nervous system disorders) | 1 (4) | 1 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (4) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 2 (4) | 7 (8)
Insomnia (Psychiatric disorders) | 1 (3) | 5 (5)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (13) | 11 (14)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 2 (3) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 1 (2)
Thrombosis (Vascular disorders) | 1 (1) | 3 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=138) | Arm B (N=142)
Blood disorder (Blood and lymphatic system disorders) | 3 (6) | 5 (7)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3) | 3 (3)
Hemoglobin decreased (Blood and lymphatic system disorders) | 53 (279) | 50 (269)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 2 (8)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphatic disorder (Blood and lymphatic system disorders) | 0 (0) | 2 (5)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2 (2) | 5 (8)
Arrhythmia (Cardiac disorders) | 3 (4) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 9 (14) | 18 (25)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 5 (7) | 4 (4)
Pericardial effusion (Cardiac disorders) | 1 (1) | 3 (4)
Premature ventricular contractions (Cardiac disorders) | 0 (0) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 9 (12) | 8 (14)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 2 (14)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (9)
Ear disorder (Ear and labyrinth disorders) | 1 (3) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (2)
External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Conjunctival disorder (Eye disorders) | 0 (0) | 1 (1)
Dry eye syndrome (Eye disorders) | 2 (3) | 3 (5)
Extraocular muscle paresis (Eye disorders) | 2 (2) | 0 (0)
Eye disorder (Eye disorders) | 1 (5) | 9 (17)
Eye pain (Eye disorders) | 0 (0) | 2 (2)
Eyelid function disorder (Eye disorders) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 11 (14) | 16 (37)
Watering eyes (Eye disorders) | 2 (4) | 3 (9)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 4 (9)
Abdominal pain (Gastrointestinal disorders) | 9 (12) | 16 (24)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 57 (142) | 51 (113)
Diarrhea (Gastrointestinal disorders) | 72 (172) | 79 (210)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 16 (48) | 24 (52)
Dysphagia (Gastrointestinal disorders) | 4 (5) | 6 (9)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 46 (86) | 41 (78)
Endoscopy large bowel abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal mucositis (Gastrointestinal disorders) | 2 (4) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric mucositis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (3) | 8 (10)
Gastrointestinal disorder (Gastrointestinal disorders) | 3 (4) | 9 (10)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Hemorrhoids (Gastrointestinal disorders) | 3 (6) | 7 (9)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 21 (31) | 17 (31)
Nausea (Gastrointestinal disorders) | 101 (325) | 108 (315)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Salivary gland disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 2 (2) | 5 (5)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 54 (98) | 46 (89)
Chest pain (General disorders) | 5 (5) | 9 (12)
Chills (General disorders) | 8 (14) | 7 (12)
Edema limbs (General disorders) | 28 (47) | 29 (85)
Fatigue (General disorders) | 124 (768) | 126 (711)
Fever (General disorders) | 10 (11) | 21 (28)
Flu-like symptoms (General disorders) | 2 (2) | 2 (2)
General symptom (General disorders) | 3 (4) | 3 (4)
Ill-defined disorder (General disorders) | 0 (0) | 2 (2)
Localized edema (General disorders) | 8 (9) | 4 (7)
Pain (General disorders) | 21 (44) | 28 (46)
Visceral edema (General disorders) | 1 (1) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 4 (5) | 4 (6)
Hypersensitivity (Immune system disorders) | 2 (9) | 4 (6)
Immune system disorder (Immune system disorders) | 1 (1) | 3 (8)
Anal infection (Infections and infestations) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 3 (3) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 1 (2)
Gingival infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 9 (11) | 12 (16)
Infectious colitis (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 2 (2)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 3 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 4 (5)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 6 (9) | 10 (11)
Skin infection (Infections and infestations) | 7 (10) | 3 (4)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 14 (18) | 13 (14)
Urinary tract infection (Infections and infestations) | 4 (5) | 7 (7)
Vaginal infection (Infections and infestations) | 2 (2) | 3 (5)
Wound infection (Infections and infestations) | 1 (1) | 2 (2)
Aortic injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (3) | 3 (10)
Dermatitis radiation (Injury, poisoning and procedural complications) | 8 (9) | 9 (9)
Fracture (Injury, poisoning and procedural complications) | 1 (6) | 1 (1)
Intraoperative breast injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pharyngeal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 3 (4) | 4 (4)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 6 (6)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 1 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Alanine aminotransferase increased (Investigations) | 27 (104) | 35 (87)
Alkaline phosphatase increased (Investigations) | 14 (44) | 12 (41)
Aspartate aminotransferase increased (Investigations) | 26 (77) | 28 (78)
Bilirubin increased (Investigations) | 0 (0) | 3 (4)
Creatinine increased (Investigations) | 2 (2) | 3 (5)
Gamma-glutamyltransferase increased (Investigations) | 2 (5) | 2 (10)
Laboratory test abnormal (Investigations) | 3 (8) | 7 (22)
Leukocyte count decreased (Investigations) | 38 (129) | 35 (149)
Lymphocyte count decreased (Investigations) | 22 (99) | 21 (103)
Neutrophil count decreased (Investigations) | 70 (147) | 75 (202)
Platelet count decreased (Investigations) | 6 (6) | 13 (30)
Weight gain (Investigations) | 10 (20) | 14 (39)
Weight loss (Investigations) | 9 (17) | 8 (21)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 27 (71) | 27 (78)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 6 (6)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (14) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 16 (52) | 22 (89)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 1 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 9 (12)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 14 (33) | 15 (32)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 2 (6)
Hyponatremia (Metabolism and nutrition disorders) | 7 (9) | 7 (14)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (21) | 21 (30)
Bone pain (Musculoskeletal and connective tissue disorders) | 11 (23) | 16 (22)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 15 (17) | 14 (19)
Fibrosis (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1)
Joint disorder (Musculoskeletal and connective tissue disorders) | 3 (5) | 3 (3)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 38 (69) | 45 (103)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (6) | 8 (8)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 (4) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 39 (107) | 48 (132)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 5 (5)
Neck soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 (36) | 18 (34)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 3 (3) | 1 (2)
Cognitive disturbance (Nervous system disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 23 (34) | 23 (35)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 40 (72) | 38 (79)
Hypoglossal nerve disorder (Nervous system disorders) | 0 (0) | 1 (3)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 1 (3)
Memory impairment (Nervous system disorders) | 7 (13) | 5 (5)
Mini mental status examination abnormal (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (3)
Neurological disorder NOS (Nervous system disorders) | 2 (4) | 6 (10)
Olfactory nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 11 (22) | 15 (31)
Peripheral sensory neuropathy (Nervous system disorders) | 92 (352) | 104 (436)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (3) | 1 (1)
Taste alteration (Nervous system disorders) | 10 (37) | 20 (62)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 5 (6) | 2 (2)
Anxiety (Psychiatric disorders) | 15 (62) | 23 (60)
Confusion (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 15 (42) | 19 (50)
Insomnia (Psychiatric disorders) | 30 (73) | 43 (76)
Libido decreased (Psychiatric disorders) | 1 (1) | 1 (6)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 2 (2)
Cystitis (Renal and urinary disorders) | 2 (2) | 0 (0)
Hemoglobinuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Hemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 1 (1)
Kidney pain (Renal and urinary disorders) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 4 (4)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 2 (6)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (2)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 2 (2) | 3 (4)
Breast pain (Reproductive system and breast disorders) | 28 (38) | 28 (46)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1) | 6 (8)
Lactation disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovulation pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 5 (10)
Reproductive tract disorder (Reproductive system and breast disorders) | 1 (3) | 0 (0)
Uterine hemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Vaginal discharge (Reproductive system and breast disorders) | 2 (2) | 4 (5)
Vaginal dryness (Reproductive system and breast disorders) | 4 (7) | 4 (7)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal mucositis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 16 (23)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchial hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (54) | 21 (40)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 24 (40) | 25 (50)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 8 (13) | 13 (21)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 13 (24)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 9 (11)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 11 (23) | 10 (11)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 93 (588) | 98 (579)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (11) | 4 (6)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 8 (11) | 5 (6)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 17 (26) | 15 (28)
Nail disorder (Skin and subcutaneous tissue disorders) | 33 (71) | 42 (93)
Pain of skin (Skin and subcutaneous tissue disorders) | 4 (7) | 6 (7)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (16) | 14 (14)
Rash acneiform (Skin and subcutaneous tissue disorders) | 15 (21) | 16 (29)
Rash desquamating (Skin and subcutaneous tissue disorders) | 24 (42) | 40 (59)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (6)
Skin disorder (Skin and subcutaneous tissue disorders) | 12 (22) | 9 (15)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 9 (24) | 25 (60)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (5)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Sweating (Skin and subcutaneous tissue disorders) | 7 (10) | 7 (13)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 2 (5) | 8 (10)
Hemorrhage (Vascular disorders) | 2 (2) | 4 (6)
Hot flashes (Vascular disorders) | 40 (101) | 45 (101)
Hypertension (Vascular disorders) | 25 (100) | 24 (83)
Hypotension (Vascular disorders) | 3 (6) | 6 (10)
Peripheral ischemia (Vascular disorders) | 1 (1) | 1 (1)
Phlebitis (Vascular disorders) | 2 (3) | 0 (0)
Thrombosis (Vascular disorders) | 4 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less